CLINICAL TRIAL: NCT02690558
Title: Phase II Single Arm Study of Gemcitabine and Cisplatin Plus Pembrolizumab as Neoadjuvant Therapy Prior to Radical Cystectomy in Patients With Muscle-Invasive Bladder Cancer
Brief Title: Phase 2 Study of Pembrolizumab in Combination With Gemcitabine and Cisplatin as Neoadjuvant Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1520
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: muscle-invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pembrolizumab, gemcitabine and cisplatin (Experimental): There is one arm in this study. Subjects will receive Pembrolizumab 200mg IV on day 1 in combination with cisplatin 35mg/m2 and gemcitabine 1000mg/m2 on day 1 and day 8 every 3 weeks for 4 cycles over 12 weeks.
  Interventions: Drug: pembrolizumab, gemcitabine and cisplatin

INTERVENTIONS:
Drug: pembrolizumab, gemcitabine and cisplatin — neoadjuvant administration of pembrolizumab with gemcitabine and cisplatin prior to cystectomy
  Other Names: Keytruda; MK-3475

SUMMARY:
The purpose of this study is to evaluate whether adding pembrolizumab (Keytruda) to the combination of gemcitabine and cisplatin will improve shrinkage of the tumor before having a cystectomy, for people with muscle-invasive bladder cancer (MIBC).

DETAILED DESCRIPTION:
Primary Objective To estimate the proportion of patients with pathological downstaging to <pT2 after neoadjuvant therapy with pembrolizumab in combination with gemcitabine and cisplatin in patients with MIBC

Hypothesis: The rate of pathologic downstaging to <pT2 will improve compared to historical controls

Secondary Objectives To estimate the proportion of patients with pT0 after neoadjuvant therapy with pembrolizumab when administered in combination with gemcitabine and cisplatin in patients with MIBC

Hypothesis: The rate of pathologic downstaging to pT0 will improve compared to historical controls

To estimate event free survival (EFS) Hypothesis: EFS will be improved compared to historical controls

To estimate overall survival (OS) Hypothesis: OS will be improved compared to historical controls

To estimate the proportion of patients who are alive at 3 years (OS at 3 years) Hypothesis: OS at 3 years will be improved compared to historical controls

To characterize the toxicity profile for the combination of pembrolizumab, gemcitabine, and cisplatin Hypothesis: Pembrolizumab, gemcitabine, and cisplatin will be a safe combination with acceptable toxicity rates

Exploratory Objectives To explore the association of biological markers including PD-L1 expression and immune gene expression signatures with pathological downstaging to <pT2, pT0, EFS, and OS

To explore associations between BASE47 "basal," "claudin-low," and "luminal" subtypes of MIBC and pathological downstaging to <pT2, pT0, EFS, and OS

To characterize the change in phenotype of TILs, including delineation of effector and regulatory T cells, before and after neoadjuvant treatment

To define T cell receptor (TCR) and B cell receptor (BCR) repertoire profiles that are associated with pathological downstaging to <pT2, pT0, EFS, and OS

First the participant will receive all 3 study drugs (Pembrolizumab/Keytruda, gemcitabine and cisplatin) on the first day of a 3 week "cycle". The participant will then receive cisplatin and gemcitabine on the 8th day of the cycle.

The participant will receive the study drugs for 4 cycles for a total of 12 weeks.

Participants are followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written IRB approved informed consent and be able to follow protocol requirements.
* Be greater than or equal to 18 years of age on day of signing informed consent.
* Has a performance status of 0 or 1 on the ECOG Performance Scale
* Has histologically confirmed urothelial carcinoma of the bladder; those with mixed histology, including a component of urothelial carcinoma, are eligible. Pure small cell carcinoma, pure adenocarcinoma, and pure squamous cell carcinoma are excluded.
* Has clinical stage T2-T4a N0/X M0 urothelial carcinoma. Clinical T stage is based on the pre-study standard of care transurethral resection of the bladder tumor (TURBT) sample and imaging studies.
* Has staging scans with abdominal/pelvic CT or MRI scan and CT scan or x-ray of the chest within 4 weeks prior to treatment initiation
* Be a medically appropriate candidate for radical cystectomy as determined by an attending urologist and be planning to receive cystectomy.
* Has had no prior systemic cytotoxic chemotherapy for urothelial carcinoma (prior intravesicular chemotherapies are permitted)
* Patients must have tumor tissue from transurethral resection of the bladder tumor (TURBT) available for submission that is sufficient for correlative testing, and agree to submission of a paraffin block or 20 formalin-fixed paraffin embedded (FFPE) slides of 5-10 microns in thickness. Patients must also agree to submission of tissue from cystectomy.
* Demonstrate adequate organ function as defined in the table below; all screening labs should be performed within 10 days of treatment initiation.

Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculated creatinine clearance (CrCL; GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (Creatinine clearance should be calculated per CKD-EPI equation.) Hepatic Serum total bilirubin ≤ 1.5 X ULN (≤ 3 X ULN if Gilbert's Syndrome) OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy. If subject receiving anticoagulants, PT or PTT should be within therapeutic range of intended use of anticoagulants

* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of pembrolizumab.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from the screening visit and continue throughout the study period up to 120 days after the last dose of study therapy.

The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Life expectancy greater than 3 months
* Consents to whole blood collection prior to initiating therapy and at cystectomy for support of correlative research studies

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject meets any of the following:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of pembrolizumab.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. NOTE: see exception to use of systemic steroid as prophylactic anti-emetic prior to cisplatin in section 4.2.2. Inhaled and topical steroids are allowed.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  • Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has received prior radiation therapy to the bladder for the purpose of treating urothelial carcinoma
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has clinically relevant hearing impairment > Grade 2
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew I Milowsky, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - North Carolina Cancer Hospital (UNC), Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose TL, Harrison MR, Deal AM, Ramalingam S, Whang YE, Brower B, Dunn M, Osterman CK, Heiling HM, Bjurlin MA, Smith AB, Nielsen ME, Tan HJ, Wallen E, Woods ME, George D, Zhang T, Drier A, Kim WY, Milowsky MI. Phase II Study of Gemcitabine and Split-Dose Cisplatin Plus Pembrolizumab as Neoadjuvant Therapy Before Radical Cystectomy in Patients With Muscle-Invasive Bladder Cancer. J Clin Oncol. 2021 Oct 1;39(28):3140-3148. doi: 10.1200/JCO.21.01003. Epub 2021 Aug 24. PMID 34428076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two cancer centers between May 2016 and March 2020.
Pre-assignment Details: Of the 47 participants screened, 8 were determined to be ineligible and a total of 39 were enrolled.
Period: Overall Study
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 7
  Former smoker | 26
  Never smoker | 6
Clinical Tumor (T) stage [Count of Participants; unit: Participants] — Anatomic stage using the American Joint Committee on Cancer (AJCC) system, which is based on the size of primary tumor (T) and whether it has grown into nearby areas. Higher numbers mean the cancer is more advanced.
  Participants
    T2 | 28
    T3 | 9
    T4a | 2
Previous non-muscle invasive bladder cancer [Count of Participants; unit: Participants]
  Yes | 7
  No | 31
  Unknown | 1
Previous Bacillus Calmette-Guérin Therapy [Count of Participants; unit: Participants]
  Yes | 5
  No | 34
Eastern Cooperative Oncology Group performance status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS is a 0-5 point scale to describe a patient's level of functioning in terms of selfcare ability and activity level (lower score means higher functioning) 0-Fully active
  1. Restricted in strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory, capable of all selfcare but unable to carry out any work; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; can't carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 28
    1 | 11
Histology [Count of Participants; unit: Participants]
  Pure urothelial | 28
  Urothelial with squamous cell | 7
  Urothelial with micropapillary | 1
  Urothelial with sarcomatoid | 1
  Urothelial with signet ring | 1
  Urothelial with glandular and squamous | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Reach Pathological Downstaging (Response) at the Time of Cystectomy
Description: Pathologic (p) anatomic stage for bladder cancer uses the American Joint Committee on Cancer (AJCC) Tumor/Nodes/Metastasis (TNM) system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced.
  Pathologic staging is based on the operative and pathology report from cystectomy at the local site. A pathologic response or downstaging is defined as a reduction in stage to below pathological tumor stage 2 (<pT2) (pT0-T1N0M0)
Time Frame: 14 weeks of treatment plus cystectomy within 70 days after treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 39
percentage of patients with response | 56 [40 to 72]

2. Secondary Outcome: Percentage of Subjects That Reach Complete Pathologic Response (pT0) at the Time of Cystectomy
Description: Pathologic (p) anatomic response for bladder cancer uses the American Joint Committee on Cancer (AJCC) TNM staging system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis) (M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced.
  Pathologic staging is based on the operative and pathology report from cystectomy at the local site.
  Complete pathologic response (pT0) is defined as pT0 N0 M0.
Time Frame: 14 weeks of treatment plus cystectomy within 70 days of treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 39
percentage of patients with response | 36 [21 to 53]

3. Secondary Outcome: Event Free Survival
Description: defined from D1 of neoadjuvant treatment until progression (in those who progress prior to surgery) or until recurrence (post-surgery) or until death as a result of any cause.
Time Frame: 14 weeks of treatment plus 5 years of followup
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: OS at 3 years is defined from D1 of treatment until 3 years or death as a result of any cause
Time Frame: 14 weeks of treatment plus 3 years or until death
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Safety and toxicity will be characterized according to the reported adverse event (AE) profile using NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0, a descriptive terminology. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 14 weeks of treatment plus 30 days for toxicity followup
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 39
Participants
  Grade 1 or higher (Any toxicity) | 39
  Grade 3 or higher | 29

ADVERSE EVENTS:
Time Frame: 14 weeks of treatment plus cystectomy within 70 days after treatment plus 30 days for toxicity follow up (a total of approximately 28 weeks)
Arm/Group | Pembrolizumab, Gemcitabine and Cisplatin
All-Cause Mortality (participants affected / at risk) | 9/39
Serious Adverse Events (participants affected / at risk) | 23/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab, Gemcitabine and Cisplatin (N=39)
Acute kidney injury (Renal and urinary disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Ejection fraction decreased (Investigations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Gastrointestinal disorders - Other, specify- hematochezia (Gastrointestinal disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify pyelonephritis (Infections and infestations) | 1
Infusion site extravasation (General disorders) | 1
Injury, poisoning and procedural complications - Other, specify neobladder leak (Injury, poisoning and procedural complications) | 1
Kidney infection (Infections and infestations) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify- new cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Neutrophil count decreased (Investigations) | 3
Peripheral ischemia (Vascular disorders) | 1
Platelet count decreased (Investigations) | 5
Sepsis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Stroke (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab, Gemcitabine and Cisplatin (N=39)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Anemia (Blood and lymphatic system disorders) | 27
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Cardiac troponin I increased (Investigations) | 1
Catheter related infection (Infections and infestations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Investigations) | 11
Cystitis noninfective (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 7
Dry eye (Eye disorders) | 1
Dysgeusia (Nervous system disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Edema limbs (General disorders) | 6
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 2
Fatigue (General disorders) | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Flu like symptoms (General disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hyperthyroidism (Endocrine disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 27
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Infusion site extravasation (General disorders) | 3
Insomnia (Psychiatric disorders) | 2
Investigations - Other, specify (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 9
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 19
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Investigations) | 23
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5
Phlebitis (Vascular disorders) | 3
Platelet count decreased (Investigations) | 26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Infections and infestations) | 1
Rectal pain (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 2
Superficial thrombophlebitis (Vascular disorders) | 5
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 8
Upper respiratory infection (Infections and infestations) | 3
Urinary frequency (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 5
Urostomy obstruction (Injury, poisoning and procedural complications) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 26
Wound complication (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT02690558/Prot_SAP_000.pdf